CLINICAL TRIAL: NCT05760495
Title: Analysis of Oxidative Stress Biomarkers and Their Determinants in ART-experienced PLWH
Acronym: 4477
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4477
Record Dates: First submitted 2023-02-02; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: ART-experienced PLWH
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood sampling for evaluation of oxidative stress markers

SUMMARY:
The project aims to assess the level of oxidative stress biomarkers in HIV patients on effective antiretroviral treatment in correlation with other therapeutic, clinical, and viro- immunological parameters. The analysis aims to better characterize the patient on treatment through an innovative approach based on two specific tests for complementary assessment of total oxidant and anti-oxidant plasma capacity.

ELIGIBILITY:
Inclusion Criteria:

* ART-treated PLWH
* HIV-1 RNA< 50 copies/mL
* Stable ART therapy (at least 48 weeks)
* Signature of informed consent for study participation

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aviremic, HIV outpatients on long-term ART
Sampling Method: Non-Probability Sample
Enrollment: 543 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the levels of total oxidant and antioxidant plasma capacity | 1 year
  Quantify the levels of total oxidant and antioxidant plasma capacity antioxidant

SECONDARY OUTCOMES:
Correlation between level of oxidative stress biomarkers and several factors | 1 year
  Evaluation of the impact of therapeutic, viro-immunologic, clinical, and demographic factors on the level of oxidative stress biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Francesca Lombardi, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No